CLINICAL TRIAL: NCT02356757
Title: Preventing Amputations by Tailored Risk-based Intervention to Optimize Therapy
Acronym: PATRIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIR 14-009
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Diabetes; Foot Ulcer
Keywords: self-care; self-monitoring; medication adherence; diet; physical activity; primary prevention
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Medication Adherence; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Behavioral Intervention (PBI) (Experimental): The PBI is a 12-month long integrated, multicomponent counseling and dermal thermometry intervention targeting foot self-care, foot self-monitoring, diet, medication and physical activity. The intervention is based on self-regulation theory, the Transtheoretical Model and
  Interventions: Behavioral: Personalized Behavioral Intervention
- Current Best Practice (CBP) (Placebo Comparator): This group will receive all the enhancements that the VA has targeted to improve foot risk in diabetes and foot care, and will also receive counseling regarding preventing general health conditions.
  Interventions: Behavioral: Current Best Practice

INTERVENTIONS:
Behavioral: Personalized Behavioral Intervention — The PBI is based on self-regulation theory, the Transtheoretical Model and Prospect Theory, and will be delivered using Motivational Interviewing principles and the teach-back method. Participants will receive monthly calls targeting foot self-care, foot self-monitoring, diet, medication and physical activity for 6 months. Call/mailing frequency during the next 6 months will depend on adherence level to foot self-care and self-monitoring at 6 months.
  Other Names: PBI
  Arms: Personalized Behavioral Intervention (PBI)
Behavioral: Current Best Practice — CBP will include monthly calls from a counselor focusing on preventing conditions like colorectal cancer, flu, insomnia, vision problems, memory loss and oral disease for the first 6 months. Frequency of calls and mailings from counselors during the next 6 months will be determined by level of adherence to preventive strategies during the first 6 months.
  Other Names: CBP
  Arms: Current Best Practice (CBP)

SUMMARY:
The PATRIOT study will evaluate a risk-based personalized behavioral intervention to improve foot self-care, self-monitoring, and modifiable risks for amputation such as blood glucose, blood pressure and cholesterol in order to prevent diabetic foot ulcers in patients at higher than normal risk for amputation. This novel intervention aims to improve self-care and early detection of foot abnormalities in at-risk patients with diabetes and poor foot self-care using advanced behavioral approaches to target adherence to multiple health behaviors, including foot self-care, self-monitoring, medication adherence, dietary adherence, and physical activity simultaneously. If this promising behavioral theory-driven approach delivered using common technology (phone) to the patient at home can work in a setting where improvements in foot care are so urgent, it will be an important scientific contribution.

DETAILED DESCRIPTION:
Amputation is a devastating complication of diabetes that is preceded in > 80% of cases by foot ulcers. Veterans with diabetes are at risk for incident foot ulcers, particularly if they have neuropathy, vascular disease or anatomic abnormalities. This risk is worsened if they have poor foot self-care, poor foot self-monitoring and/or poor control of A1c and other risk factors. It is important to activate at-risk Veterans to improve self-care and self-monitoring, and lower other amputation risks.

The PATRIOT study is a randomized controlled trial (RCT) testing the effectiveness of a personalized behavioral intervention (PBI) aimed to improve foot self-care, foot self-monitoring, and modifiable risks for amputation such as A1c, BP, LDL and smoking using behavioral counseling combined with dermal thermometry. The primary specific aim is to evaluate the effect of PBI on the proportion of foot lesions (ulcerative or non-ulcerative) compared to current best practice (CBP) care for diabetes. The secondary specific aims are to evaluate the impact of PBI on foot self-care skills, foot education and adherence, A1c, BP and LDL, and quality of life at 6 months as well as its longer-term effects at 12 months; and cost-effectiveness compared to CBP. The will also examine the effect of PBI and CBP on demonstrated foot self-care, plantar pressures, inflammation, satisfaction and intervention acceptability.

The investigators will randomize 404 adults with diabetes who are at higher than normal risk of foot ulcers [Risk score of 1, 2 or 3 (with no history of ulcers or amputations)] to the PBI and CBP equally. The PBI is a cohesive, personalized intervention targeting foot self-care and self-monitoring that includes dermal thermometry, diet, exercise, and medication-taking incorporating self-regulatory theory, the Transtheoretical Model and Prospect Theory and delivered using Motivational Interviewing principles and the teach back method. The interventions will be standardized and fidelity of the intervention will be maintained. Through a blinded RCT, the investigators will test the effect of PBI in relation to CBP. Key outcomes are non-ulcerative and ulcerative lesions, foot-care skills, foot care education, adherence to diet and medication, general and foot health-specific quality of life, A1c, BP, and LDL. Outcomes will be measured at baseline, 6 and 12 months. All analyses will be intent-to-treat.

This study will evaluate a cohesive risk-stratified personalized behavioral intervention aimed to improve self-care, enhance self-monitoring and reduce incident ulcers in adults without a previous diabetic foot ulcer. This study applies established behavioral theories combined with new technology to intervene and improve care for adults with diabetes who are at risk for amputation. If this promising theory-driven primary prevention approach to prevent foot lesions can work in a clinical setting where improvements in foot care are urgently needed, it will be an important scientific contribution that could lower the risk of amputation in adults with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diabetes and PAVE score 1, 2 or 3, drug therapy for > 6 months
* An available phone
* At least 2 primary care visits in the previous 1.5 years at the recruitment site

Exclusion Criteria:

* Patients with acute CVD events < 3 months ago
* 86 poor estimated short-term survival (< 1 year)
* Recent major surgery (< 3 months)
* Inability to exercise
* Prior toe or foot amputation
* Prior foot ulcer
* Temporary residence in the area
* Inability to provide consent will be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Ulcerative and non-ulcerative Foot lesions | 12 months
  High-resolution standard view digital photographs of the feet and footwear will be obtained and reviewed by the investigators blinded to group assignment, and a suspected ulcer or nonulcerative plantar lesion below the malleoli will be referred to a blinded (as to group assignment) adjudicators, all clinical experts. Lesions will be judged as absent/nonulcerative lesion/ulcer

SECONDARY OUTCOMES:
Foot care skills | 12 months
  The investigators will use the Veterans foot self-care education and behavior survey to assess foot care.
Foot-care education | 12 months
  The investigators will use the Veterans foot self-care education and behavior survey to assess basic foot-care education and extended foot-care education. This survey was developed and validated in high-risk Veterans.
Medication adherence | 12 months
  This will be assessed primarily by refill frequency using the pharmacy database , supplemented by the self-reported medication-taking scale. Refill compliance is an objective measurement of medication adherence that utilizes pharmacy records to assess the proportion of time a patient has medication available.
Diet | 12 months
  Diet will be assessed by food frequency questionnaire
Physical activity | 12 months
  Physical activity will be assessed via accelerometer.
A1c | 12 months
  Fasting blood will be processed for A1c.
Systolic blood pressure | 12 months
  Blood pressure will be measured with an Omron automated machine and the mean of 6 BP's over 2 hours. used.
LDL | 12 months
  Fasting blood will be processed for LDL cholesterol.
Health-related quality of life | 12 months
  General health-related quality of life will be assessed using the Veterans SF-12. The investigators will also measure foot health-specific quality of life. Measures are reliable and valid.
Cost-effectiveness | 12 months
  The investigators will measure direct medical costs (costs of drugs, tests, supplies, personnel, and facilities),direct non-medical costs (transportation), and indirect (patient's time and caregiver's time). The investigators will also calculate quality-adjusted life years using the ED-5D survey to adjust for health states.

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD MSc, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No